CLINICAL TRIAL: NCT03310060
Title: Reducing Blood Loss During Total Knee Arthroplasty Using Tisseel: A Prospective Randomized Control Trial
Brief Title: Reducing Blood Loss Using Tisseel in TKA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 201700271A3
Record Dates: First submitted 2017-10-02; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Total Blood Loss
MeSH Terms: conditions — Exsanguination | interventions — Fibrin Tissue Adhesive; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tisseel combined Tranexamic acid (Active Comparator): Drug: Tisseel® Applied on potential bleeding sites. The entire content was 4 mL.
  Drug: Tranexamic acid Intravenous application of tranexamic acid 15mg/kg before surgical incision and 3 hours after surgery
  Interventions: Drug: Tisseel; Drug: Tranexamic Acid
- Tranexamic acid (Placebo Comparator): Drug: Tranexamic acid Intravenous application of tranexamic acid 15mg/kg before surgical incision and 3 hours after surgery
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tisseel — Tisseel® (Fibrin Sealant, 4ml, Baxter) was applied on potential bleeding sites: the femoral insertion of the posterior cruciate ligament, the lateral genicular artery after resection of the meniscus, the posterior capsule of the knee joint, the bony surfaces not covered by the implant as well as the pinholes (femur and tibia). The entire content of a 4 mL vial containing the active product was used
  Other Names: Fibrin Sealant
  Arms: Tisseel combined Tranexamic acid
Drug: Tranexamic Acid — Drug: Tranexamic acid Intravenous application of tranexamic acid 15mg/kg in 100 ml normal saline before surgical incision and 3 hours after surgery
  Other Names: Transamin

SUMMARY:
The purpose of this study is to conduct a prospective randomized controlled trial to investigate the blood-conservation effect of the topical hemostatic agents in patients receiving primary TKA procedures. The investigators will also observe if there is increased risk of blood transfusion rate by using topical hemostatic agents or not.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is associated with considerable blood loss and increasing needs for allogenic blood transfusion. Previous studies demonstrated a transfusion rates ranging from 6% to 38% after standard TKAs. Transfusion carries significant risks of cardiopulmonary embarrassment, disease transmission, immunological reaction and postoperative infection.

The major causes of postoperative blood loss following TKA are attributed to surgery itself which induces a considerable activation of the coagulation cascade and local fibrinolysis, the latter is further enhanced after release of the tourniquet at the end of surgery. Tranexamic acid (TXA), an inhibitor of fibrinolysis, was reportedly effective reducing blood loss after standard TKA. Previous experiences in minimally invasive (MIS) TKA showed that intraoperative infusion of TXA reduced 45% of postoperative blood loss and needs for transfusion from 20% to 4%. However, the safety to use TXA systemically in TKAs especially in high risk patients remains controversial. A recent study by Nishihara et al. demonstrated that use of TXA in total hip arthroplasty did not appear to affect the prevalence of either proximal DVT or PE. Another study by Xie J et al. also showed the incidence of postoperative VTE was unchanged when TXA was administered in primary unilateral TKA, but in their study the total occurrence of vascular occlusive events was statistically significantly higher (17.55% Vs 9.35%, p < 0.001) in the TXA group. However, in this two studies the patient with high risk of thromboembolic events (ischemic heart disease, chronic renal failure on hemodialysis, cerebral infarction, previous VTE disease, thrombophilia associated with genetic diseases) were excluded.

The investigators believe the use of hemostatic agent topically in patients with high risk of thromboembolism can avoid its systematic effect and decrease its potential perioperative risk of thromboembolic complications (arterial thrombosis, myocardial infarction and pulmonary embolism). On the other hand, thrombin-based hemostatic agents, Tisseel®, have been widely used in surgical procedure including gynecology, general surgery, and orthopedics which were still attracting the attention and interest of multitudinous surgeons. Some recent studies demonstrated that topic use of Tisseel® in primary TKA can reduce hemoglobin decline and calculated total blood loss after TKA and is not related to adverse reactions or complications such as wound infection, venous thromboembolism events(VTE). But there were another studies showed Tisseel® does not reduce blood loss in TKA procedures.

The purpose of this study therefore is to conduct a prospective randomized controlled trial to investigate the blood-conservation effect of the topic hemostatic agents and their safety in a primary TKA procedures in patients with risk of thromboembolic events. The first group by topical Tisseel and intravenous TXA application, and the second group of placebo IV TXA then observe whether there is difference in the blood-conservation effect by total blood loss calculation, hemoglobin loss and transfusion requirement among different groups.

ELIGIBILITY:
Inclusion Criteria:

* After cardiologist or neurologist's evaluation, patients who was classified as low-risk of perioperative risk with advanced knee osteoarthritis who was failure of medical treatment or rehabilitation and within age limit

Exclusion Criteria:

* Preoperative Hemoglobin ≦12 g/dl History of infection or intraarticular fracture of the affective knee, Renal function deficiency (GFR < 30 ml/min/1.73m2), Elevated liver enzyme, history of liver cirrhosis, impaired liver function and coagulopathy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Total blood loss after operation | from the operation to the postoperative day 3
  Total blood loss was calculated according to Nadler et al., which used maximum postoperative reduction of the Hb level adjust for weight and height of the patient. The formula is as follows, Total blood loss = (Total blood volume x [change in Hb level / preoperative Hb level])x1000+volume transfused

SECONDARY OUTCOMES:
Incidence of any thrombotic events | within 30 days of the operation
  the composite of any suspected venous thromboembolism events, ischemic heart diseases, or cerebrovascular accidents
Incidence of wound infection after surgery | within 30 days of the operation
  composite of wound poor healing, superficial wound infection, and deep infection requiring return to surgery
Blood transfusion requirement | from the operation to postoperative day 14
  compare blood transfusion requirement between two groups
Calculated blood loss from drainage | from the operation to the postoperative day 2 until drainage removal
  blood loss was calculated according to the hemovac drainage record every eight hours after operation until removal.